CLINICAL TRIAL: NCT02222844
Title: Improving Radical Treatment Through MRI Evaluation of Pelvic Sigmoid Cancers
Acronym: IMPRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Pelican Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DOCUMAS: 23HH8201
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Colorectal Neoplasms; Colon, Sigmoid; Magnetic Resonance Imaging; General Surgery
Keywords: Cancer; Colorectal Neoplasms; Colon, Sigmoid; Magnetic Resonance Imaging; General Surgery; Postoperative Complications
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Preoperative CT scan (No Intervention): CT-imaging of chest and abdomen / pelvis before surgery (standard treatment)
- Preoperative MRI scan (Experimental): Standard treatment plus an additional MRI scan before surgery
  Interventions: Other: Preoperative MRI scan
- Observational (No Intervention): Observational only

INTERVENTIONS:
Other: Preoperative MRI scan — Standard preoperative CT of abdomen, chest and pelvis plus interventional preoperative MRI scan.
  Arms: Preoperative MRI scan

SUMMARY:
Patients with suspected or proven sigmoid colon adenocarcinoma, eligible for curative treatment whose MRI can be reviewed prior to surgery and has no decision regarding radical treatment are eligible. Patient are randomised to the control arm which the standard care of preoperative CT imaging and subsequent discussion by the Multidisciplinary Team or the interventional arm which has the additional use of MRI imaging and subsequent discussion by the Multidisciplinary Team. Patients are followed up at 1 and 3 years together with QoL questionnaires.

DETAILED DESCRIPTION:
A randomised phase II multicentre trial, IMPRESS will determine whether the use of MRI imaging in staging sigmoid cancers results in a change to the treatment plan by identifying more high risk tumours compared to those patients who were staged using CT imaging. The proposed intervention will be additional radiological and pathological assessment and the reporting of supplementary diagnostic information which would not otherwise have been available. This may affect treatment according to local MDT protocols and also affect the provision of prognostic information to patients in subsequent discussions.

ELIGIBILITY:
Inclusion Criteria:

1. Have a suspected or proven sigmoid colon adenocarcinoma
2. Is eligible for curative treatment
3. Has no irresectable metastatic disease
4. MRI can be reviewed by an MDT prior to surgery
5. Has no decision regarding radical treatment
6. Have provided written informed consent to participate in the study
7. Be aged 16 years or over

Exclusion Criteria:

1. Have metastatic disease (including resectable liver metastases)
2. Have a synchronous second malignancy
3. Are contraindicated for MRI
4. Are contraindicated for or have allergy to Buscopan (e.g. glaucoma, small or large bowel obstruction, GFR<30)
5. Have severe co-morbidities or previous medical history that prevent the application of eventual chemo/radiotherapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Observational Phase: To measure the difference in staging of sigmoid cancer on CT and MRI. | 3 years after last recruit
  Direct comparison of proportion of patients staged as high and low risk for recurrence between CT vs MRI findings
Randomised Phase: To measure the difference in treatment stratification policy caused by the difference in staging on CT and MRI. | 3 years after last recruit
  Direct comparison of proportion of patients undergoing preoperative treatment or extended surgery between patients staged with CT vs MRI

SECONDARY OUTCOMES:
To compare the recurrence rates of sigmoid tumours staged by CT and MRI according to predicted prognostic risk. | 3 years after last recruit
  Comparison of proportion of recurrences in patients staged as low vs high risk on CT vs MRI
To compare disease free survival of patients staged by CT and MRI according to predicted prognostic risk. | 1 and 3 years after last recruit
  Kaplan-Meier curves of disease free survival in patients staged as low vs high risk on CT vs MRI
To compare the quality of surgery by pathology of patients staged by CT and MRI according to predicted prognostic risk. | 5 years
  Grade of specimen using pathology TNM8 stratified by TNM8 staging on CT vs MRI
To compare CRM positivity rates on pathology of patients staged by CT and MRI according to predicted prognostic risk | 3 years after last recruit
  CRM positivity rates on pathology in patients staged as low vs high risk on CT vs MRI
To compare baseline and post-treatment stage on imaging against pathology and clinical outcomes of patients staged by CT and MRI. | 3 years after last recruit
  Comparison of proportion of patients staged as low vs high risk on CT vs MRI with pathology high and low risk and against outcomes
To compare perioperative morbidity and mortality of patients staged by CT and MRI according to predicted prognostic risk. | 3 years after last recruit
  Comparison of perioperative morbidity of patients stratified by preoperative treatment between patients staged with CT vs MRI
To compare quality of life of patients staged by CT and MRI according to predicted prognostic risk. | 1 and 3 years after last recruit
  Comparison of quality of life between patients staged with CT vs MRI by questionnaire (EORTC QLQ-CR29)
To compare permanent defunctioning stoma rates in patients staged by CT and MRI according to predicted prognostic risk. | 3 years after last recruit
  Comparison of proportion of stomas not reversed within 3 years postoperative follow-up in patients staged with CT vs MRI

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, Principal Investigator — Imperial College London
Locations (16):
- United Kingdom (16):
  - Hinchingbrooke Hospital, Huntingdon, Cambridgeshire
  - Leighton Hospital, Crewe, Cheshire
  - University Hospital of North Tees, Stockton-on-Tees, County Durham
  - Croydon University Hospital, Thornton Heath, Croydon
  - Chesterfield Royal, Chesterfield, Derbyshire
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - St Mark's Hospital, Middlesex, Harrow
  - Maidstone Hospital, Maidstone, Kent
  - Queen Elizabeth the Queen Mother Hospital, Margate, Kent
  - North Manchester General Hospital, Crumpsall, Manchester
  - University Hospital of South Manchester & Manchester Royal Infirmary, Wythenshawe, Manchester
  - Harrogate District Hospital, Harrogate, North Yorkshire
  - Musgrove Park Hospital, Taunton, Somerset
  - Yeovil District Hospital, Yeovil, Somerset
  - Royal Marsden Hospital, Sutton, Surrey
  - Salisbury District Hospital, Salisbury, Whiltshire